CLINICAL TRIAL: NCT04956770
Title: STIMO-PARKINSON: Study on Feasibility of Targeted Epidural Spinal Stimulation (TESS) to Improve Mobility in Patients With Parkinson's Disease
Brief Title: Study on Feasibility of Targeted Epidural Spinal Stimulation (TESS) to Improve Mobility in Patients With Parkinson's Disease
Acronym: STIMO-PARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jocelyne Bloch (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor-Investigator, Jocelyne Bloch, Professor, Neurosurgeon, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STIMO-PARK2021
Record Dates: First submitted 2021-05-31; First posted 2021-07-09 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Spinal Cord Stimulation System; DBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single center, non-randomized, interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation supported by TESS (Experimental): Patient will be asked to come to the hospital for three types of patient sessions:
  * Stimulation configuration sessions: TESS protocols will be setup and optimized during this phase.
  Duration: minimum 4 sessions over 2 weeks, maximum 20 sessions over a month. In addition, some sessions at a free frequency as needed during rehabilitation will be programed (maximum once a week).
  * TESS-supported rehabilitation sessions: Patients will undergo an in-clinic rehabilitation training regime supported by TESS.
  Duration: 24 sessions spread over minimum three months and maximum five months
  * Pre- and post-rehabilitation evaluation sessions: four clinical evaluation sessions will take place focusing on assessment of locomotion, balance and PD related deficits.
  Interventions: Procedure: Implantation surgery

INTERVENTIONS:
Procedure: Implantation surgery — The intervention involves the implantation of:
  * a neurostimulator: the Activa® RC from Medtronic
  * a stimulation electrode paddle array: the Specify™ SureScan® 5-6-5 from Medtronic

SUMMARY:
The purpose of the STIMO-PARKINSON study is to evaluate the safety and preliminary efficacy of Targeted Epidural Spinal Stimulation (TESS) system to induce modulation in leg muscle recruitment in patients with advanced Parkinson's disease, and its capacity to improve key gait and balance deficits when employed in the context of a rehabilitation process of 3 to 5 months.

DETAILED DESCRIPTION:
The study intervention consists of 7 phases preceded by pre-screening:

* enrolment and eligibility
* baseline
* surgery
* main phase of the study
* home-use
* end of main study phase
* (optional and conditional): 3 years follow-up

At baseline, general information and Parkinson related medical history are collected. Clinical evaluations are also completed without and with current therapy, (i.e. NO(MED+DBS), and MED+DBS conditions). Finally, quality of life questionnaires are collected for the patient as well as expectations questionnaires for the physiotherapists involved in the study.

The main phase of the study consists of:

* Stimulation configuration sessions during which TESS protocols will be setup and optimized. This procedure aims to configure the spatial and temporal parameters of TESS that will recruit specific muscle groups. Specific TESS protocols will be configured for various motor tasks which will be used during the rehabilitation phase and clinical evaluations.
* TESS-supported rehabilitation sessions during which patients will undergo an in-clinic rehabilitation training regime supported by TESS.
* Evaluation sessions during which four clinical evaluation sessions will take place focusing on assessment of locomotion, balance and PD related deficits. The tests will be done when patients are:

  (i) in NO(MED+DBS) condition (without any therapy, i.e. without medication and DBS OFF) (ii) in MED+DBS condition (the patient's standard therapeutical condition, i.e. usual medication dose and DBS ON) (iii) in TESS+MED condition (usual medication dose, TESS ON, DBS OFF) (iv) in TESS+MED+DBS condition (usual medication dose, TESS ON, DBS ON)

Participants are allowed to use the investigational system independently if deemed safe and beneficial as assessed by the Principal Investigator (Home-Use Phase).

One year after patient enrolment, the patient will come for follow up visits where he will again perform an evaluation session for each therapy condition as described above, to evaluate the long-term evolution.

If the therapy has been safe and beneficial, they can extend their study participation by entering the Follow-Up period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease with III-IV Hoehn-Yahr stage, exhibiting severe gait difficulties and postural instability
* With Medtronic DBS implant and receiving medication for Parkinson's disease
* Aged 18 to 80 years
* Stable medical, physical and psychological condition as considered by the Investigators in accordance with treating physician and treating neurologist.
* Must agree to comply in good faith with all conditions of the study and to attend all required study training and visit
* Must provide and sign the study's Informed Consent prior to any study-related procedures

Exclusion Criteria:

* Severe or chronic medical disorder pre-existing PD diagnosis affecting rehabilitation
* Active oncological disease requiring heavy treatments and frequent MRI controls
* Having an implanted device that is active (e.g., pacemaker, implantable cardiac defibrillator) whose interference with the investigational system's neurostimulator (Activa RC) is not confirmed safe by the CE-mark of the device, or having an indication that might lead to implantation of such device
* Inability to follow study procedures, e.g. due to language problems, psychological disorders, dementia as considered by the Investigators in accordance with treating physician and treating neurologist
* Hematological disorders with an increased risk of hemorrhagic event during surgical interventions
* Life expectancy of less than 12 months
* Pregnant or breast feeding
* Participation in another interventional study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Occurence of all SAEs and AEs deemed or related to study procedure or to the study investigational system | Through study completion, an average of 6 months
  Evaluate the safety of TESS at supporting locomotor rehabilitation in patients with Parkinson's Disease

SECONDARY OUTCOMES:
EMG measurements of muscle recruitment in response to stimulation of increasing amplitudes for different contact configurations | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy outcome of TESS to induce modulations in muscle recruitment selectivity by measuring the EMG response to iterative stimulation pulses of increasing amplitude for different contact configurations
Maximum voluntary contraction (MVC) of single joints | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy of TESS on motor performance through changes in single joint leg muscle strength and fatigue
Muscle Fatigue Test | At baseline and during the 5-month TESS-supported rehabilitation phase
  Measure the time the patient can maintain a certain percentage of his MVC measured in the MED+DBS condition. This is used to assess the preliminary efficacy of TESS on motor performance through changes in single joint leg muscle strength and fatigue
10-meter walk test | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy of TESS on motor performance through changes in gait speed and endurance
6 minute walk test | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy of TESS on motor performance through changes in gait speed and endurance
Timed up and Go test and its cognitive version, as custom-made FOG circuit | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy of TESS for alleviating deficits specific to PD related to freezing of gait (FOG)
Kinematic analysis | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy of TESS for alleviating deficits specific to PD related to posture using motion sensors acquisition system
Mini Balance Evaluation Systems Test (mini-BESTest) | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy of TESS for alleviating deficits specific to PD related to balance
Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess the preliminary efficacy of TESS for alleviating deficits specific to PD related to motor and non-motor functions. Higher scores indicate greater impact of Parkinson's disease symptoms

OTHER OUTCOMES:
Cortical (EEG) and subcortical signals (LFP from the subthalamic nucleus) | At baseline and during the 5-month TESS-supported rehabilitation phase
  Assess changes in brain activity patterns induced by TESS-supported physical training to get insight into the effects of TESS on brain dynamics. This will be done in the four therapy conditions for rest, for single-joint leg tasks and, if results are encouraging, for gait
Quality of life questionnaire PDQ-39 | At baseline and during the 5-month TESS-supported rehabilitation phase
  Evaluate the effect of TESS-supported rehabilitation on quality of life of patients through the Parkinson's Disease Questionnaire (PDQ-39). The score ranges from 0 to 100, lower scores reflect better quality of life
Quality of life questionnaire ABC-Q | At baseline and during the 5-month TESS-supported rehabilitation phase
  Evaluate the effect of TESS-supported rehabilitation on quality of life of patients through the Activities-specific Balance Confidence Scale (ABC-Q). The score ranges from 0% to 100%, higher score reflects higher level of physical functioning
Quality of life questionnaire FOG-Q | At baseline and during the 5-month TESS-supported rehabilitation phase
  Evaluate the effect of TESS-supported rehabilitation on quality of life of patients through the Freezing of Gait Questionnaire (FOG-Q). The score ranges from 0 to 24, higher scores correspond to more severe FOG
Quality of life questionnaire KPPS | At baseline and during the 5-month TESS-supported rehabilitation phase
  Evaluate the effect of TESS-supported rehabilitation on quality of life of patients through King's Parkinson's disease pain scale. The score ranges from 0 to 168, higher scores correspond to higher pain.
Therapist expectations and learnings questionnaire | At baseline (before the patient is implanted) and at the time of study completion
  Obtain information concerning the perceived efficacy of TESS-supported rehabilitation for Parkinson's patients and whether they would recommend tis new therapy for general clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strauss I, Kalia SK, Lozano AM. Where are we with surgical therapies for Parkinson's disease? Parkinsonism Relat Disord. 2014 Jan;20 Suppl 1:S187-91. doi: 10.1016/S1353-8020(13)70044-0. PMID 24262178
- [Background] Courtine G, Bloch J. Defining ecological strategies in neuroprosthetics. Neuron. 2015 Apr 8;86(1):29-33. doi: 10.1016/j.neuron.2015.02.039. PMID 25856483
- [Background] Courtine G, Gerasimenko Y, van den Brand R, Yew A, Musienko P, Zhong H, Song B, Ao Y, Ichiyama RM, Lavrov I, Roy RR, Sofroniew MV, Edgerton VR. Transformation of nonfunctional spinal circuits into functional states after the loss of brain input. Nat Neurosci. 2009 Oct;12(10):1333-42. doi: 10.1038/nn.2401. Epub 2009 Sep 20. PMID 19767747
- [Background] Capogrosso M, Milekovic T, Borton D, Wagner F, Moraud EM, Mignardot JB, Buse N, Gandar J, Barraud Q, Xing D, Rey E, Duis S, Jianzhong Y, Ko WK, Li Q, Detemple P, Denison T, Micera S, Bezard E, Bloch J, Courtine G. A brain-spine interface alleviating gait deficits after spinal cord injury in primates. Nature. 2016 Nov 10;539(7628):284-288. doi: 10.1038/nature20118. PMID 27830790
- [Background] Fuentes R, Petersson P, Siesser WB, Caron MG, Nicolelis MA. Spinal cord stimulation restores locomotion in animal models of Parkinson's disease. Science. 2009 Mar 20;323(5921):1578-82. doi: 10.1126/science.1164901. PMID 19299613
- [Background] Yadav AP, Nicolelis MAL. Electrical stimulation of the dorsal columns of the spinal cord for Parkinson's disease. Mov Disord. 2017 Jun;32(6):820-832. doi: 10.1002/mds.27033. Epub 2017 May 12. PMID 28497877
- [Background] Santana MB, Halje P, Simplicio H, Richter U, Freire MAM, Petersson P, Fuentes R, Nicolelis MAL. Spinal cord stimulation alleviates motor deficits in a primate model of Parkinson disease. Neuron. 2014 Nov 19;84(4):716-722. doi: 10.1016/j.neuron.2014.08.061. Epub 2014 Oct 30. PMID 25447740
- [Background] Cai Y, Reddy RD, Varshney V, Chakravarthy KV. Spinal cord stimulation in Parkinson's disease: a review of the preclinical and clinical data and future prospects. Bioelectron Med. 2020 Mar 16;6:5. doi: 10.1186/s42234-020-00041-9. eCollection 2020. PMID 32232113
- [Background] Prasad S, Aguirre-Padilla DH, Poon YY, Kalsi-Ryan S, Lozano AM, Fasano A. Spinal Cord Stimulation for Very Advanced Parkinson's Disease: A 1-Year Prospective Trial. Mov Disord. 2020 Jun;35(6):1082-1083. doi: 10.1002/mds.28065. Epub 2020 Apr 20. No abstract available. PMID 32311155
- [Background] Cury RG, Carra RB, Capato TTC, Teixeira MJ, Barbosa ER. Spinal Cord Stimulation for Parkinson's Disease: Dynamic Habituation as a Mechanism of Failure? Mov Disord. 2020 Oct;35(10):1882-1883. doi: 10.1002/mds.28271. No abstract available. PMID 33068473